CLINICAL TRIAL: NCT01209481
Title: Impact of Educational Group Intervention on the Consumption of Fruit and Vegetables by Adult People Attended to Primary Health Care.
Brief Title: Impact of Educational Group Intervention on the Consumption of Fruit and Vegetables
Acronym: fvphc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Maria Antonieta de Barros Leite Carvalhaes, São Paulo State University - Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: upeclin/HC/FMB-Unesp-48
Record Dates: First submitted 2010-08-30; First posted 2010-09-27 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Inclusion Criteria:; Adult; No Pregnancy; No Lactation; No Morbidity
Keywords: fruits; vegetables; primary health care; nutritional education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional education (Experimental)
  Interventions: Behavioral: nutritional education group action
- control (No Intervention)

INTERVENTIONS:
Behavioral: nutritional education group action — The educational group activities will consist of two-hour group dynamics and cooking workshops once a week and for five weeks.
  Arms: Nutritional education

SUMMARY:
The right to food and nutrition is established in the Universal Declaration of Human Rights as they are basic requirements for promoting and protecting good health. They can also be instruments to evaluate the quality of life of human beings and communities. Awareness of a healthy diet is the first step in behavioral change, and nutritional education can be an instrument for avoiding diseases resulting from both intake deficit and excess. Educational group actions can change food intake. This study will aim at evaluating, planning and implementing the impact of a nutritional education group action concerning the consumption of fruit and vegetables in adult and elderly individuals attended to by a Primary Health Care (PHCU) Unit. It will be a randomized assay involving two groups comprising male and females individuals distributed in the following fashion: Intervention Group, in which the educational group action (EGA) will be performed in addition to routine activities; and Control Group, the individuals from which will only participate in the routine activities in the PHCA (Teaching Health Care Unit). The total sample will comprise 80 individuals with 40 in each group. In order to determine the consumption of fruit and vegetables, a weekday and a Sunday 24-hour recalls will be performed 2 (short-term effects) and 6 (medium-term effects) months after completing the intervention. The educational group activities will consist of two-hour group dynamics and cooking workshops once a week and for five weeks. Serum carotenoid dosages will also be performed in the two groups by sub-sampling (n=40) with the purpose to validate the estimated intake of fruit and vegetables obtained from the recalls.

ELIGIBILITY:
Inclusion Criteria:

* adult healthy

Exclusion Criteria:

* pregnancy, lactation, morbidity

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
consumption of fruit and vegetables | Jan 2011

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonieta BL Carvalhaes, PHD, Principal Investigator — Sao Paulo State University, Faculty of Medicine
Locations (1):
- Sao Paulo State University, Faculty of Medicine, Botucatu, São Paulo, Brazil